CLINICAL TRIAL: NCT04771689
Title: Assess the Efficacy of Buprenorphine/Naloxone Micro-Dosing for Postoperative Pain Management in Opioid-Tolerant Patients
Brief Title: Buprenorphine/Naloxone Micro-Dosing for Postoperative Pain Management in Opioid-Tolerant Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi Zhang, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000553
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Post-operative Pain
Keywords: pain; pain management
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine/Naloxone (Active Comparator): Subjects will take a maximum dose of 4 mg buprenorphine and 1 mg naloxone with concurrent administration of other intravenous or oral opioids needed.
  Interventions: Drug: Buprenorphine/Naloxone
- Standard Medication Regiment (No Intervention): Subjects will take conventional intravenous or oral opioid management.

INTERVENTIONS:
Drug: Buprenorphine/Naloxone — Subjects will be randomized into one of the treatment groups and will follow the assigned medication schedule for the length of their hospital stay, at least 6 days.
  Other Names: Suboxone
  Arms: Buprenorphine/Naloxone

SUMMARY:
A randomized clinical study evaluating the effect of buprenorphine/naloxone (bup/nx) sublingual film on postoperative pain management in opioid-tolerant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Opioid tolerance, defined as the daily use of greater than or equal to 60mg of oral morphine or an equianalgesic dose of any other opioid for more than 7 days immediately prior to the surgery
2. Undergoing orthopedic or general surgery
3. 18 years of age or older
4. Willing and able to adhere to the study protocol and follow-up schedule
5. Able to provide written informed consent to participate in the clinical trial
6. If female and of childbearing potential, agree to use an effective method of birth control approved by the study investigators throughout the study

Exclusion Criteria:

1. Buprenorphine or buprenorphine/naloxone use in the last two weeks
2. Patients receiving pre-, intra-, or post-operative regional blocks or neuraxial anesthesia
3. Patients receiving postoperative ketamine or lidocaine boluses or infusions
4. Patients receiving postoperative nonsteroidal anti-inflammatory drugs (NSAIDs) for pain control
5. Diagnosis of severe medical or psychiatric conditions contraindicated for bup/nx treatment
6. Liver disease, including clinically significant transaminitis, active hepatitis infection, cirrhosis with evidence of impaired synthetic function
7. Anticipated deterioration of health due to discontinuation of medications that are contraindicated with bup/nx
8. Positive pregnancy test for women of childbearing potential
9. Known allergy or sensitivity to bup/nx
10. Anticipation that the subject may need to initiate pharmacological treatment during the trial that is deemed unsafe by the study physician or could prevent study completion
11. Current participation in additional pharmacologic research study
12. Active suicidal ideation as determined by PI or study clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores | through study completion, an average of 6 days
  To examine changes in pain scores daily from the day of surgery to the hospital discharge day.
Postoperative Opioid Consumption | through study completion, an average of 6 days
  To compare opioid consumption after surgery between the buprenorphine/naloxone group and the standard medication regiment group.
Length of Hospital Stay | through study completion, an average of 6 days
  To compare the length of hospital stay after surgery between the buprenorphine/naloxone group and the standard medication regiment group.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Karina de Sousa, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared with other researchers in the future.

REFERENCES:
- See also: Massachusetts General Hospital Center for Translational Pain Research — http://www.massgeneral.org/translationalpainresearch/